CLINICAL TRIAL: NCT05965063
Title: Evaluation of the Influence of Bifidobacterium on the Infants With Food Allergic
Brief Title: The Role of Bifidobacterium Intervention in Food Allergic Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BifidobacteriumRJH
Record Dates: First submitted 2023-06-24; First posted 2023-07-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Food Allergy in Infants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary avoidance for allergy food (Other): strict avoidance of the specific allergenic food
  Interventions: Other: allergy food avoidance
- bifidobacterium intervention (Experimental): Bifidobacterium M-16V for 12 weeks while strictly avoidance of the specific allergenic food
  Interventions: Dietary Supplement: Bifidobacterium M-16V
- Healthy control (No Intervention): without intervention

INTERVENTIONS:
Dietary Supplement: Bifidobacterium M-16V — Bifidobacterium M-16V was dosed at 10 billion colony forming unit (CFU) (equal to 6 drops)/day for 12 weeks.
  Arms: bifidobacterium intervention
Other: allergy food avoidance — strict avoidance of the specific allergenic food
  Arms: Dietary avoidance for allergy food

SUMMARY:
Infant food protein allergy is the most common allergic disease in children, which can lead to infantile-specific dermatitis, intestinal inflammation, and so on. Dietary avoidance is a common strategy for food protein allergy in infants and young children. However, the hidden etiology of food protein allergy or multiple food allergies often leads to poor efficacy. The aim of this study is to observe the clinical effectiveness of Bifidobacterium intervention on food allergy.

ELIGIBILITY:
Inclusion Criteria:

* 0 -12 months infant
* Infants that are allergic (confirmed by an allergist) to at least one of the main food allergens (cow's milk, egg, soy or wheat) and is following an elimination diet to at least one of these allergens.

Exclusion Criteria:

* Patients had used probiotics within 1 month prior to the study
* Allergy or intolerance to probiotics or their excipient
* Serious primary diseases of the cardiovascular, nervous, respiratory,hepatobiliary immunology，and endocrine systems;

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
The milk related symptom score at the 4th week | Treatment for 4-week
  Compare the clinical symptoms of infants at the 4th week by milk-related symptom score (0-33) and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The milk related symptom score at the 8th week | Treatment for 8-week
  Compare the clinical symptoms of infants at the 8th week by milk-related symptom score (0-33) and higher scores mean a worse outcome.
The milk related symptom score at 12th week | Treatment for 12-week
  Compare the clinical symptoms of infants at the 12th week by milk-related symptom score (0-33) and higher scores mean a worse outcome.

OTHER OUTCOMES:
The percentile number of height at the 4th, 8th and12th week | Treatment for 4-week, 8-week and 12-week
  Compare the Percentile number of height of infants at the 4th, 8th and 12th week
The percentile number of weight at the 4th, 8th and 12th week | Treatment for 4-week, 8-week and 12-week
  Compare the Percentile number of weight of infants at the 4th, 8th and 12th week
The percentile number of head circumference at the 4th, 8th and 12th week | Treatment for 4-week, 8-week and 12-week
  Compare the Percentile number of head circumference of infants at the 4th, 8th and 12th week
The composition of intestinal microbiome | Treatment for 4-week, 8-week and 12-week
  All subjects faeces will be collected and analyzed by high-throughput metagenomic sequencing to find the characteristics and composition of intestinal microbiome at the 4th, 8th and 12th week to analyze the intestinal microbiome composition
The composition of intestinal microbiome metabolites | Treatment for 4-week, 8-week and 12-week
  This will be detected and analyzed by liquid chromatography-mass spectrometry (LC-MC) non-targeted metabolomics at the 4th, 8th and 12th week to analyze the intestinal microbiome metabolites.
the messenger ribonucleic acid (mRNA) expression of blood | Treatment for 12-week
  The mRNA expression of blood will be detected and analyzed by blood RNA-seq at the 12th week

CONTACTS AND LOCATIONS:
Overall Officials: CHUNDI Xu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No